CLINICAL TRIAL: NCT04582110
Title: Retinal and Choriocapillaris Vascular Features in Patients With Beta Thalassemia by Means of Optical Coherence Tomography Angiography
Brief Title: The Role of OCTA in Patients Affected by Beta Thalassemia
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 1002/19
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Beta Thalassemia: Patients with previous diagnosis of Beta Thalassemia
  Interventions: Diagnostic Test: Optical coherence tomography angiography
- Control Group: Healthy fellow eyes without actual and previous ocular trauma
  Interventions: Diagnostic Test: Optical coherence tomography angiography

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography angiography — Each subject underwent Optical coherence tomography angiography (a non-invasive, fast, diagnostic imaging technique)

SUMMARY:
To investigate, using optical coherence tomography angiography (OCTA), the retinal and choriocapillaris vascular features in patients affected by Beta Thalassemia. Moreover we analyzed the structural retinal parameters (ganglion cell complex and retinal nerve fiber layer), using optical coherence tomography (OCT) in these patients

DETAILED DESCRIPTION:
Beta Thalassemia is one of the most common genetic hemoglobinopathy characterized by a defective β globulin chain synthesis leading to hemolysis and ineffective erythropoiesis.

The study investigated the changes in retinal and choriocapillaris vascular features using optical coherence tomography angiography, a novel and noninvasive diagnostic technique that allows a detailed analysis of retinal and choriocapillaris blood flow.

ELIGIBILITY:
Inclusion Criteria:

* age older than 35 years
* diagnosis of Beta Thalassemia
* absence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* absence of significant lens opacities, low-quality OCT and OCT-A images.

Exclusion Criteria:

* age older than 50 years
* absence of diagnosis of Beta Thalassemia
* presence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* presence of significant lens opacities, low-quality OCT and OCT-A images.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participans were older than 35 years with diagnosis of Beta Thalassemia. They did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal and choriocapillaris features in patients with Beta Thalassemia, using optical coherence tomography angiography. | Four months
  The parameters analyzed by optical coherence tomography angiography were: retinal and choriocapillaris vessel density

SECONDARY OUTCOMES:
The measurements of retinal structural parameters in patients with Beta Thalassemia, using optical coherence tomography. | Four months
  The parameters analyzed by optical coherence tomography were: ganglion cell complex and retinal nerve fiber layer

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples "Federico II", Naples, Italy